CLINICAL TRIAL: NCT03465657
Title: Sodium Sources and Sodium Intake in a Representative Sample of Spanish Children and Its Effects on Body Weight and Blood Pressure
Brief Title: Sodium Sources and Sodium Intake in a Representative Sample of Spanish Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Rosa María Ortega Anta, Full Professor, Universidad Complutense de Madrid
Other Study IDs: PR6/13-18866
Record Dates: First submitted 2018-03-06; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Urinary Sodium Excretion; Salt Intakes; Body Weight
Keywords: Child Health; Sodium intake; Food Sources; Blood Pressure; BMI; Urinary sodium excretion
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The 24-h urine sample were collected and kept for future analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous evidence shows that sodium intake in Spanish adult population is over the recommended limits and this high sodium intake is related with difficulties in body weight control and blood pressure control.

The aim of this study is to stablish a direct relationship between salt intake and the health parameters previously mentioned in a representative sample of Spanish schoolchildren between 7-11 years old. The investigators are applying a 3-day dietary records to collect dietary data, and collecting 24-h urine samples in order to analyse biochemical indicators of sodium intake and other nutrients. Anthropometric data are also being recorded and body composition is also analysed using bioimpedance technique.

DETAILED DESCRIPTION:
Specific Aims

1. To stablish the average sodium intake in Spanish children, using a 24-h urine sample and validated dietary questionnaires.
2. To compare 24-hour urinary sodium measurement to the dietary survey method
3. To study the relationship between sodium intake and blood pressure levels in Spanish scholars.
4. To analyze the relationship between sodium intake and overweight/obesity in Spanish children using anthropometric and bioimpedance analysis measures.
5. To identify main food sources of sodium in the diet of Spanish schoolchildren and the use of discretionary salt.
6. Provide new data for monitoring sodium intake in Spanish schoolchildren and design campaigns to reduce their intake.
7. To provide reference data of sodium intake on a representative sample of the Spanish child population for European and international databases.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 11 years old

Exclusion Criteria:

* Those who have any clinical problem, which may modify the results of the analysis: metabolic or chronic diseases (liver, kidney, diabetes, hypothesis or hyperkalemia), pharmacological treatment during the 3 months prior to the study with corticosteroids, insulin, diuretics or other drugs that may modify blood pressure figures, surgery or serious infectious diseases in the previous 6 months.
* Those who were not in the school when the measures were taken.

Ages: 7 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: Representative population of Spanish Children between 7-11 years old from schools of different regional communities.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-10-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
24-h urinary sodium excretion in Spanish schoolchildren | Through study completion, an average of 2 years
  Estimation of salt intake by 24 h urinary sodium excretion

SECONDARY OUTCOMES:
Common sodium food sources | Through study completion, an average of 2 years
  Quantify the contribution of different foods to the total sodium intake

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Ortega Anta, Full Prof., Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Dto. Nutrición y Ciencia de los Alimentos (NUTRYCIAL). Facultad de Farmacia. UCM, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aparicio A, Rodriguez-Rodriguez E, Cuadrado-Soto E, Navia B, Lopez-Sobaler AM, Ortega RM. Estimation of salt intake assessed by urinary excretion of sodium over 24 h in Spanish subjects aged 7-11 years. Eur J Nutr. 2017 Feb;56(1):171-178. doi: 10.1007/s00394-015-1067-y. Epub 2015 Oct 19. PMID 26482149